CLINICAL TRIAL: NCT07405632
Title: The Impact of Supplementation With Hericium Erinaceus (Lion's Mane) Extract on Cognitive Functioning: A Double-blind Placebo-controlled Study
Brief Title: The Impact of Supplementation With Hericium Erinaceus (Lion's Mane) Extract on Cognitive Functioning
Acronym: HECOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: Omyu Sp. z o.o. (Unknown); SWPS University Doctoral School (Unknown)
Responsible Party: Principal Investigator, Maria Kossowska, Msc, University of Social Sciences and Humanities, Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Hericium erinaceus - Cognition; GW2 (Other Grant/Funding Number: SWPS University Doctoral School)
Record Dates: First submitted 2026-01-26; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Attention; Memory; Cognitive Function and Well-Being
Keywords: Lion's Mane; Hericium erinaceus; Cognitive functioning; Attention; Well-being

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, and placebo-controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hericium erinaceu (Experimental): This is a group of participants who will receive Hericium erinaceu during the duration of the study.
  Interventions: Dietary Supplement: Hericium erinaceus Supplementation
- Placebo (Placebo Comparator): This is a group of participants who will receive placebo during the wole duration of the study.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hericium erinaceus Supplementation — Each participant will take extract from the fruiting bodies of Lion's Mane mushroom (Hericium erinaceus; trade name: Lion's Mane Focus; manufacturer: Omyu sp. z o.o., Warsaw, Poland). Composition: mineral water, food-grade ethanol <22%, dried Lion's Mane fruiting bodies 20,000 mg. * Dosage: 1ml per day*. * Instructions: Take before 1:00 PM.*
  Arms: Hericium erinaceu
Dietary Supplement: Placebo — Each participant will take placebo. Composition: mineral water, food-grade ethanol <22%, caramel food flavouring 0.2%. * Dosage: 1ml per day*. * Instructions: Take before 1:00 PM.*
  Arms: Placebo

SUMMARY:
The goal of this study is to determine whether supplementation with Hericium erinaceus (Lion's Mane) extract enhances selected cognitive functions in healthy, actively working, middle-aged women. We aim to investigate a broad spectrum of cognitive functions to identify which, if any, are affected both immediately and after prolonged supplementation with Hericium erinaceus extract.

Our main research questions are as follows:

1. Can Hericium erinaceus extract supplementation modify cognitive status?
2. Is there an immediate effect on cognition following a single intake of Hericium erinaceus extract?
3. Does prolonged supplementation with Hericium erinaceus extract influence cognitive functioning?
4. Which cognitive functions are affected, and will the patterns differ between immediate effects and those observed after long-term supplementation?
5. Will participants report subjective cognitive enhancement?

Our main hypotheses are as follows:

1. A single dose of Hericium erinaceus extract will produce an acute effect, improving attention 45 minutes after intake.
2. An eight-week supplementation period with Hericium erinaceus extract will produce a chronic effect, improving long-term memory.
3. The investigators will compare Hericium erinaceus extract with a placebo (a visually identical substance that contains no active ingredients) to determine whether the extract effectively enhances cognitive functioning.

Participants will:

1. Take a Hericium erinaceus extract or placebo capsule daily for 2 months.
2. Visit SWPS University for baseline assessments before beginning supplementation (T0), a follow-up assessment 45 minutes after the initial intake (T1), and additional assessments at 1 week (T2) and 2 months (T3).
3. Complete neuropsychological testing and questionnaires during the T1, T2, and T3 visits.
4. Maintain their usual dietary habits throughout the study.

ELIGIBILITY:
Inclusion Criteria:

- residing in Warsaw, Poland or the surrounding area.

Exclusion Criteria:

* pregnancy or lactation,
* history of head injury with neurological consequences,
* history of neurological disorders or diseases,
* chronic use of antibiotics,
* use of antibiotics within the last 30 days,
* chronic use of antifungal medications,
* use of antifungal medications within the last 30 days,
* allergies or intolerance to mushrooms (especially Lion's Mane),
* consumption of caffeinated beverages (e.g., coffee, energy drinks) prior to the study visit.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 85 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-10-11 (Actual); Study Completion 2025-10-11 (Actual)

PRIMARY OUTCOMES:
Change in d' score in old/new recognition test (ONR) to assess long-term memory | 45 minutes after the first dose, and at 1 week and 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  The old/new word recognition task is designed to assess episodic memory. It is consisted of two phases: a learning phase and a recognition phase. During the learning phase, participants viewed 30 pictures on the computer. In the recognition phase, participants were presented with 30 "old" and 30 "new" pictures in random order and were asked to determine whether each picture had been shown during the learning phase. To analyze episodic memory task we followed Macmillan and Creelman (2005) signal detection theory, where d' is the ability to discriminate between signal and noise (between old and new stimuli), H stands for the proportion of correct changes detected (hit rate), and F stands for the proportion of changes incorrectly reported (false alarm rate). d' = zH - zF
Change in Differentiation score in California Verbal Learning Test (CVLT) to assess long-term memory | 45 minutes after the first dose, and at 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  California Verbal Learning Test (CVLT) measure the verbal learning and memory. It measures how well individuals learn and recall verbal material, assessing both short-term and long-term memory. The Differentiation score measures the ability to distinguish between correct and incorrect responses. Scores range from 0 to 16, with higher scores indicating better outcome.
Change in Concentration score in d2 Test of Attention (d2-R) - to assess attention | 45 minutes after the first dose, and at 8 week after the start of supplementation with Hericium erinaceus extract or placebo.
  Scores range from 0 to 308, with higher scores indicating better outcome.
Change in the number of correctly marked target characters in the d2 Test of Attention (d2-R) - to assess attention. | 45 minutes after the first dose, and at 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  Scores range from 0 to 308, with higher scores indicating better outcome.
Change in cueing effect in the Posner Cueing Task to assess attentional orienting efficiency | 45 minutes after the first dose, and at 1 week and 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  The Posner Cueing Task assesses visuospatial selective attention, specifically the speed and efficiency of orienting attention to a cued location. To analyze this efficiency, we calculated the cueing effect. This is defined as the difference in mean reaction time between invalidly cued trials and validly cued trials (RT invalid-RT valid). A larger cueing effect indicates a higher "cost" of disengaging attention from an incorrect location and shifting it to the correct target.
Change in reaction time to validly cued targets in the Posner Cueing Task to assess attentional orienting speed | 45 minutes after the first dose, and at 1 week and 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  The Posner Cueing Task assesses visuospatial selective attention, specifically the speed and efficiency of orienting attention to a cued location. To assess attentional orienting speed, the primary outcome is the reaction time to the target in valid trials (where the cue correctly predicts the target location). A shorter reaction time indicates faster attentional orienting to the predicted spatial location. Reaction times are measured in milliseconds.

SECONDARY OUTCOMES:
Changes in Beck Depression Inventory (BDI) total score to assess symptoms of depression | 45 minutes after the first dose, and at 1 week and 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  Scores range from 0 to 63, with higher scores indicating more severe depressive symptoms.
Changes in the Fatigue Assessment Scale (FAS) total score to assess symptoms of chronic fatigue | 45 minutes after the first dose, and at 1 week and 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  Scores range from 10 to 50, with higher scores indicating greater fatigue.
Change in Color Trails Test (CTT) completion time - CTT1 to assess several attention and executive functions especially perceptual tracking, sustained and divided attention | 45 minutes after the first dose, and at 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  A maximum time limit of 240 seconds (4 minutes) is applied.
Change in Color Trails Test (CTT) completion time - CTT2 to assess several attention and executive functions especially perceptual tracking, sustained and divided attention | 45 minutes after the first dose, and at 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  A maximum time limit of 240 seconds (4 minutes) is applied.
Change in Wechsler Adult Intelligence Scale (WAIS) Digit Span Forward subset total score to assess short-term auditory memory | Baseline (prior to intervention), 45 minutes after the first dose, and at 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  Scores range from 0 to 14, with higher scores indicating better outcome.
Change in Wechsler Adult Intelligence Scale (WAIS) Digit Span Backward subset total score to assess short-term auditory memory | Baseline (prior to intervention), 45 minutes after the first dose, and at 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  Scores range from 0 to 14, with higher scores indicating better outcome.
Change in Wechsler Adult Intelligence Scale (WAIS) Digit Symbol Substitution subtest total score to assess cognitive processing speed, visual-motor coordination, and sustained attention | Baseline (prior to intervention), 45 minutes after the first dose, and at 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  Scores range from 0 to 39, with higher scores indicating better outcome.
Changes in Memory Functioning Questionnaire (MFQ) total score | 45 minutes after the first dose, and at 1 week and 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  The Memory Functioning Questionnaire (MFQ) is a self-report instrument designed to assess subjective memory functioning and memory complaints. We utilized the version developed by Gilewski et al. (1990), which consists of 64 items divided into four main subscales: Frequency of Forgetting, Seriousness of Forgetting, Retrospective Functioning, and Mnemonics Usage. Higher scores on the MFQ indicate a higher level of perceived memory functioning.
Change in Operation Span (OSPAN) capacity load to assess working memory capacity | 45 minutes after the first dose, and at 1 week and 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  The Operation Span (OSPAN) task is a standard measure of working memory capacity, requiring participants to solve mathematical equations while simultaneously remembering a sequence of letters. The primary outcome measure is the capacity load, which represents the sum of all letters from sets that were recalled perfectly in their correct order. A higher capacity load score indicates a greater ability to maintain and manipulate information in the face of distraction, reflecting superior working memory capacity.
Change in energy scores | Baseline (prior to intervention), 45 minutes after the first dose, and at 1 week and 8 weeks after the start of supplementation with Hericium erinaceus extract or placebo.
  Scores range from 0 to 100, with higher scores indicating higher subjective energy at the time of assessment.

OTHER OUTCOMES:
Score in the Raven's Progressive Matrices test | 45 minutes after the first dose of supplementation with Hericium erinaceus extract or placebo.
  The Raven's Progressive Matrices test is used to measure the level of general intelligence, understood as fluid intelligence. It is scored on a scale from 0 to 60, with higher scores indicating better outcome.
Score in Adherence to the Mediterranean diet | 45 minutes after the first dose of supplementation with Hericium erinaceus extract or placebo.
  The scale ranges from 0 to 7, with higher scores reflecting greater adherence to the Mediterranean diet.

CONTACTS AND LOCATIONS:
Locations (1):
- SWPS University, Warsaw, Masovian Voivodeship, Poland